CLINICAL TRIAL: NCT03894306
Title: Understanding How Medication is Stored in the Home
Status: Withdrawn | Type: Observational
Why Stopped: Unable to enroll any patients due to COVID
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-01297
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Poisoning
MeSH Terms: conditions — Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- medication lock box + brief counseling
  Interventions: Other: Medication lock box; Other: brief counseling
- medication lock bag + brief counseling
  Interventions: Other: medication lock bag; Other: brief counseling
- brief counseling alone
  Interventions: Other: brief counseling

INTERVENTIONS:
Other: Medication lock box — given a lock box and instructed on how to use the device.
  Groups: medication lock box + brief counseling
Other: medication lock bag — given a lock bag and instructed on how to use the device.
  Groups: medication lock bag + brief counseling
Other: brief counseling — After completing the per-intervention survey, a research assistant or investigator will perform brief counseling, including educational handouts and information on safe medication storage

SUMMARY:
The goal of this study is to increase safe medication storage practices in homes with young children in order to prevent unintentional childhood poisonings.

As a step toward meeting this goal, this study aims to determine if an intervention to promote safe storage to patients who have young children in their home, including provision of a lock box or lock bag along with brief counseling versus brief counseling alone, results in 1) increased locked storage (and overall safe medication storage practices) of high-risk prescription medications in the home; 2) increased safe medication storage practices of other medications in the home; and 3) improved safe medication storage related knowledge and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the buprenorphine clinic, high A1c clinic, or palliative care clinic at NYC Health + Hospitals/Bellevue
* Patient prescribed at least one high-risk mediation. A high-risk medication defined as a prescription medication that may cause significant toxicity or death with the ingestion of only one pill or a single adult dose.
* A child less than six years old is present in the patient's home on average at least 8 hours per week.

Exclusion Criteria:

* Inability to speak and read English or Spanish
* No phone number for follow-up or unwilling to do follow-up by phone or in person
* Prior enrollment
* Patient was involved in pilot study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in the buprenorphine clinic, high A1c clinic, or palliative care clinics at NYC Health + Hospitals/Bellevue who are prescribed at least one high-risk medication and have a child less than six years old present in his/her home on average at least 8 hours per week.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with locked storage of all high-risk prescription medications at one month follow-up. | 1 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Su, MD, Principal Investigator — NYU Langone Health - Toxicology